CLINICAL TRIAL: NCT03756909
Title: The Effect of Neutrophil Lymphocyte Ratio and Platelet Lymphocyte Ratio on Intraoperative and Postoperative Complications in Pediatric Patients Undergoing Otolaryngology
Brief Title: Effect of Neutrophil Lymphocyte-platelet Lymphocyte Ratio on Complications in Pediatric Patients
Acronym: NLOPEDI
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Asist.Prof. MD, Aydin Adnan Menderes University
Other Study IDs: NLOPEDİ
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia; Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adenoidectomy group: Operations of adenoidectomy
- adenotonsillectomy group: Operations of adenotonsillectomy

SUMMARY:
The aim of this study was to investigate the relationship between NLR, PLR and postoperative complications in children undergoing adenotonsillectomy and adenoidectomy.

DETAILED DESCRIPTION:
Between the dates of February 1, 2018 and June 30, 2018, patients between 2-10 years of age, ASA I-II, elective adenotonsillectomy and adenoidectomy under general anesthesia were planned to be included in the study. The number of neutrophils, lymphocytes and platelets will be taken from the hospital registry system taken preoperatively and the NLR and PLR ratios will be calculated.

All patients in the operating room will be started with routine monitoring and anesthesia. Hemodynamic data during surgery will be recorded. The entrance to the operating room (T1), 5 minutes after the start of anesthesia (T5), 15 minutes (T15), 30 minutes (T30) and 45 minutes (T45) will be recorded in the follow-up form of the anesthesia. The fasting period of the patients and the drugs and fluids applied during surgery will be recorded from the anesthesia form. At the end of the operation, the patients who were taken to the recovery room at the end of the surgery will be evaluated with 1 point, 15 minutes, 30 minutes, 1 hour and 4 hours and 6 hours vomiting using the 4 point nausea scale.

Introduction to recovery room using Modified Eastern Ontario Children's Hospital Pain Scale (mCHEOPS), postoperative pain at 15 min, 30 min, 1 hr and 4 hr. Analgesic requirement will be recorded. Bronchospasm, agitation, etc. will be recorded by evaluating whether there are complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective adenotonsillectomy and adenoidectomy under general anesthesia

Exclusion Criteria:

* Immunodeficiency
* Children of parents who do not want to participate in the study
* Use of anticoagulants
* Children with hematological disease

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 2-10 years
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The effect on postoperative complications of neutrophil lymphocyte ratio in adenotonsillectomy and adenoidectomy PAIN | Postoperative 6 hours
  Pain level will be evaluated by using CHEOPS (Children's Hospital of Eastern Ontario Pain Scale ) pain score. The scale includes six categories of pain behavior (Cry, facial, verbal, torso, touch, and legs). A score ranging from 0 to 2 or 1 to 3 is assigned to each activity and the total score ranges between 4 and 13.
The effect on postoperative complications of neutrophil lymphocyte ratio in adenotonsillectomy and/or adenoidectomy POVN | Postoperative 6 hours
  Pain level will be evaluated by using POVN score. Evaluation of nausea and vomiting was performed by a four-point scale; 0: No nausea and/or vomiting, 1: mild nausea and/or vomiting which does not require treatment, 2: nausea and/or vomiting requiring treatment and 3: vomiting resistant to antiemetic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)